CLINICAL TRIAL: NCT03340259
Title: Proximal Remnant Intestinal Colonization in Newborn Infants With Enterostomy: a Longitudinal Study
Brief Title: Intestinal Colonization in Newborn Infants With Enterostomy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universidade do Porto (Other)
Collaborators: CINTESIS - Center for Health Technology and Services Research, Porto (Unknown); Hospital Dona Estefânia, Centro Hospitalar de Lisboa Central, Lisboa (Unknown); Universidade Nova de Lisboa (Other)
Responsible Party: Sponsor
Other Study IDs: MICROENTE_01
Record Dates: First submitted 2017-11-08; First posted 2017-11-13 (Actual); Last update posted 2017-11-13 (Actual); Status verified 2017-07

CONDITIONS: Newborn Infants With Enterostomy by Congenital Malformations of the Gastrointestinal Tract, Necrotizing Enterocolitis and Spontaneous Intestinal Perforation
Keywords: Congenital malformations of the gastrointestinal tract; Enterostomy; Microbiota; Necrotizing enterocolitis; Newborn Infants; Spontaneous intestinal perforation
MeSH Terms: conditions — Enterocolitis, Necrotizing

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Enterostomy effluent
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Newborn infants with enterostomy: Infants with enterostomy after surgery due to congenital malformations of the gastrointestinal tract, necrotizing enterocolitis, and spontaneous intestinal perforation
  Interventions: Procedure: Exposure(s) of interest: enterostomy

INTERVENTIONS:
Procedure: Exposure(s) of interest: enterostomy — Newborn infants with congenital malformations of the gastrointestinal tract, necrotizing enterocolitis, and spontaneous intestinal perforation commonly require surgery and enterostomy. In these infants samples of the enterostomy effluent will be collected and DNA extracted for microbiota identification.

SUMMARY:
The human microbiota, a collection of microorganisms mostly settled in the gastrointestinal tract, plays a major role in the maintenance of the hosts' health and in development of disease as well. Exposure to different conditions early in life contributes to distinct "pioneer" bacterial communities, which shape the newborn infants' development and influence their later physiological, immunological and neurological homeostasis. Newborn infants with congenital malformations of the gastrointestinal tract (CMGIT), necrotizing enterocolitis (NEC), and spontaneous intestinal perforation (SIP) commonly require abdominal surgery and enterostomy. While intestinal microbiota has been extensively studied in infants with anatomically uninterrupted intestine, the knowledge of longitudinal intestinal colonization in this population is scarce.

This is an exploratory, observational, and longitudinal prospective study, primarily aimed to determine longitudinally the colonization of the proximal remnant intestine, in newborn infants with enterostomy after surgery (three weeks) for CMGIT, NEC and SIP. The secondary aim is to explore the associations of the colonization with the mode of delivery, gestational age, postnatal age, duration of fasting, type of enteric feeding, antimicrobial therapy, H2-receptor antagonist therapy, and length of proximal remnant intestine.

ELIGIBILITY:
Inclusion criteria: newborn infants with enterostomy after surgery for CMGIT, NEC or SIP, consecutively admitted

Exclusion criteria: newborn infants with diagnosed inborn errors of metabolism, those whose parents or legal guardians will not consent to participate or withdrawn the consent, and those who had not complete 21 days of follow-up.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Newborn infants with enterostomy after surgery for CMGIT, NEC or SIP recruited at the NICU of Hospital Dona Estefânia, Centro Hospitalar de Lisboa Central, Lisbon, Portugal.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2017-06-21 (Actual); Primary Completion 2020-06 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Pattern of postsurgical intestinal microbiota colonization specific to each underlying condition | The first sample will be collected as close as possible after placement of ostomy bag. From the first collection, new samples will be collected every 3 days, until the 21st day after surgery
  Longitudinal postsurgical microbiota colonization of the proximal remnant intestine, specific to each underlying condition

SECONDARY OUTCOMES:
Associations of types of microorganism identified with below defined clinical variables | The aforementioned clinical variables will be collected daily and the enterostomy effluent collected from the first placement of ostomy bag and every 3 days thereafter up to 21 days after surgery
  Associations of microbiota colonization with the mode of delivery, gestational age, postnatal age, duration of fasting, type of enteric feeding, antimicrobial therapy, H2-receptor antagonist therapy, and length of proximal remnant intestine.

CONTACTS AND LOCATIONS:
Overall Officials: Luís Pereira-da-Silva, MD, PhD, Principal Investigator — Hospital Dona Estefânia, Centro Hospitalar de Lisboa Central; Conceição Calhau, PhD, Principal Investigator — Universidade Nova de Lisboa
Locations (1):
- Neonatal Intensive Care Unit, Hospital Dona Estefânia, Centro Hospitalar de Lisboa Central, Lisbon, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Barreiros Mota I, Marques C, Faria A, Neto MT, Cordeiro-Ferreira G, Virella D, Pita A, Pereira-da-Silva L, Calhau C. Colonisation of the proximal intestinal remnant in newborn infants with enterostomy: a longitudinal study protocol. BMJ Open. 2019 Nov 24;9(11):e028916. doi: 10.1136/bmjopen-2019-028916. PMID 31767579